# Medical University of South Carolina CONSENT TO BE A RESEARCH SUBJECT

**TITLE OF RESEARCH:** Ketamine-assisted Motivational Enhancement Therapy for the Treatment of Tobacco Use Disorder

## **Concise Summary**

Your consent is being sought for a research study. Participation is voluntary. The purpose of the study is to examine whether an investigational medication called ketamine is able to improve treatment outcomes for smoking cessation. If you are eligible and you decide to participate in the study, your participation will last approximately 12 weeks, or 3 months.

The study will involve an initial screening visit. You will complete questionnaires and interviews in a private room. The questionnaires and interviews will be related to your physical and mental health. The initial phase of the study will involve 3 clinic visits (once per week, lasting 2-3 hours per visit). At each of these visits, you will be asked to answer several questionnaires and provide a saliva sample to test for recent nicotine use and a urine sample to check for pregnancy in persons of child-bearing potential. At the initial visit, you will be asked to provide a urine sample for a drug screen. You will meet with a study coordinator to discuss motivations and goals for smoking cessation. You will then be administered the study medication by an injection into your shoulder muscle and will be monitored by a study clinician until you feel back to your usual self. A clinician will be available during and after treatment to discuss your experience. At the clinic visits where the study medication is administered, you will not be allowed to drive home. You will also meet with our study physician 4 and 8 weeks after your final medication session. These follow-ups (lasting half hour to an hour) will include questionnaires and saliva nicotine testing and can be completed virtually (ie, via secure video software).

There are risks of participating in the study that are described in this document. The most significant risks include temporary high blood pressure, anxiety, and having the sensation that you are detached from your body or having an altered perception of time or your body. There is also a risk of loss of confidentiality, although steps will be taken to minimize this risk. Because it is not known if the study medication is safe in pregnancy, if you are of childbearing potential, you will complete a pregnancy test at each visit when medication is to be taken to be sure that you are not pregnant.

Your potential benefits from participating include having a lower desire to smoke cigarettes or feeling like it is easier to remain abstinent from cigarettes, however, personal benefits cannot be guaranteed. Your alternative is not to participate in the study. Alternative treatments are available for individuals with tobacco use disorder including medications such as varenicline, bupropion, and nicotine





## A. PURPOSE OF THE RESEARCH

You are being asked to volunteer for a research study. Research studies are voluntary and include only people who choose to take part. Please read this consent form carefully and take your time making you decision. As the study doctor or study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand.

The purpose of this study is to examine the ability of a medication called ketamine to reduce the severity of tobacco use disorder, specifically to decrease cigarette use. Ketamine is currently approved by the Food and Drug Administration (FDA) to reduce pain during some surgeries. However, ketamine is considered "investigational use" in this study, meaning that the FDA has not approved it for the treatment of tobacco use disorder. This is a Phase II study of ketamine, meaning that it has established use for other purposes and researchers are now testing this medication in larger populations. The purpose of this study is to evaluate the safety and effectiveness of ketamine in the treatment of tobacco use disorder. You are being asked to participate because you are over 21 years of age and you currently have tobacco use disorder. Approximately 8 people will take part in this study.

The investigator in charge of the study is Dr. Emily Amador at the Medical University of South Carolina (MUSC). This study is being conducted with funding from a grant from the National Institute on Drug Abuse (NIDA) through the Diversity in Addiction Research Training program.

## **B. PROCEDURES**

If you agree to be in this research study, the following will happen:

- 1. Screening and Baseline Visit (approximately 2-3 hours in length):
  - The initial visit will involve the following:
    - Completion of written questionnaires related to your mental and physical health.
       Questionnaires will also be related your previous use of other substances, such as alcohol, level of cigarette use, craving levels for nicotine, motivation to quit smoking, and other symptoms such as anxiety and insomnia.
    - An interview with a clinician about questions related to your physical and mental health.
    - A basic physical exam like what you would get at a checkup and includes blood pressure, pulse, and temperature measurements.
    - We will complete a baseline electrocardiogram (EKG). This is a test of the function of your heart and involves placing small adhesive pads with wires attached on your chest. After the adhesive pads are placed, a monitor shows a picture of the electrical activity of your heart, which is printed out on paper. This test usually takes less than 10 minutes to complete. If you have had this test done within the previous 365 days at MUSC, your medical record will be reviewed. If this test was normal, you may not have to complete.





#### Version Date: 2/28/2023

- A saliva sample will be collected at baseline and follow-up to determine recent nicotine use.
- o A urine sample to test for recent use of recreational psychoactive drugs
- A urine pregnancy test (only if you are an individual of childbearing potential). The urine pregnancy test must be negative to participate.
- After staff has reviewed all the information collected, you will be contacted to inform you of
  your eligibility status. If you are eligible to enroll and choose to continue participation, you
  will be asked to come for weekly medication visits for 3 weeks. If you are not found eligible
  and/or do not choose to continue in the study, additional community resources can be made
  available to you upon request.
- If you are an individual of childbearing potential, precautions should be taken throughout the
  course of the medication phase of the study. Examples of acceptable methods of birth control
  for participants involved in the study includes: birth control pills, patch, IUD, condom, sponge,
  diaphragm with spermicide, or avoiding sexual activity that could cause you to become
  pregnant. In addition, urine pregnancy tests will be completed at baseline visit. If you are
  pregnant, you will be withdrawn from the study.
- 2. Medication Visits (approximately 2-3 hours each in length):
  - If you are eligible and decide to participate in the study, over the next 3 weeks you will come
    to the study center once per week to complete the medication visits. You will be encouraged
    to come well hydrated, but in a fasting state (i.e. not having eaten for 2 hours prior to the
    treatment visit). At these visits, you will complete questionnaires and saliva testing much like
    the ones completed at the screening visit. These tasks will take about 30 minutes.
  - You will complete a urine pregnancy test prior to each medication session (only if you are an individual of childbearing potential). The urine pregnancy test must be negative to participate.
  - You will also be weighed prior to administration of the investigational medication to ensure accurate dosing.
  - Each medication visit will include motivational-based psychotherapy, which is a type of
    counseling that focuses on motivation and setting goals. Examples of this therapy include
    setting an intention for your session, supportive talk as needed throughout medication
    session, reflection on the experience of the session afterwards, and setting goals to work on
    after each session.
  - Prior to being administered the investigational medication, you will sit in a chair and be guided
    by the study doctor through a basic relaxation exercise. This exercise will help you to focus
    on your breathing and is designed to help reduce any anxiety you may feel related to the
    medication sessions. The relaxation exercise will last about 10 minutes.
  - After you complete the relaxation exercise, you will have your blood pressure and heart rate
    checked, and you will have a small, painless monitoring device placed on your finger which
    will measure the oxygen levels in your blood throughout the medication session.






Version Date: 2/28/2023

- The investigational medication, ketamine, is given by intramuscular injection. After receiving the injection, you will be instructed to rest in a chair. After approximately 60-90 minutes, you will take complete several short questionnaires.
- Your blood pressure will be checked again, and if it is normal, the blood oxygen finger device will be removed, and the visit will be completed. If your blood pressure is high, you are feeling anxious, or you are not feeling like yourself, you will continue to be monitored by the study doctor until these symptoms return to normal.
- After completing the visit, you will be asked to have someone drive you home. If you do not
  have someone that can drive you home and live locally, transportation (such as a taxi) will
  be provided for you at no cost to you. If you live more than 20 miles from the study site and
  cannot arrange your own transportation you will not be able to participate in this study.
  Reimbursement will be a flat rate of \$100 to cover compensation for time and travel for each
  visit.
- 3. Follow-Up Visits (approximately 30 to 60 minutes each in length):
  - Completion of written questionnaires related to your mental and physical health.
     Questionnaires will also be related to recent use of tobacco products, your cravings and
     withdrawal symptoms related to nicotine and motivation to quit smoking as well as
     symptoms of anxiety and insomnia. At these visits, you will complete saliva testing for
     recent nicotine use.
  - Follow-up visits can be completed either in person or virtually (via secure video software) depending on your preference.

### C. DURATION

Participation in the study will take about 6 visits over a period of approximately 3 months. There will be an initial screening visit (approximately 2-3 hours), 3 study medication visits (approximately 2-3 hours each), and 2 follow-up visits (approximately 30 minutes).

## D. RISKS AND DISCOMFORTS

There are risks involved with participating in this study, including risks associated with ketamine, study procedures, and loss of confidentiality.

#### Ketamine Risks:

Ketamine may cause some, all or none of the side-effects listed below. These effects are generally temporary and resolve within one hour, although they may last up to six hours. A study physician will monitor you until these symptoms resolve.

More Likely (10 percent to 50 percent):

 Perceptual changes (e.g. distortion of time and space, sense of illusions) and dissociation (including a sense of detachment or altered sense of reality)

IRB Number: «ID»
Date Approved «ApprovalDate»




## Version Date: 2/28/2023

- Feeling abnormal or drunk
- Elevated blood pressure
- Elevated heart rate
- Anxiety
- Sedation (sleepiness)
- Vertigo or dizziness
- Nausea
- Decreased pain threshold

## Less Likely (5 percent to 10 percent):

Injection site swelling, pain, redness, or discomfort

## Rare (less than or equal to 5 percent):

- Bladder discomfort or increased frequency of urination (also called cystitis)
- Anaphylaxis

#### Unknown risks:

- High amounts of ketamine given to rats caused damage to different parts of the brain. It is not known whether this finding in rats will happen in humans. The amount of ketamine given to the rats was higher than what you will receive in this study.
- The added effect of repeated ketamine infusions is unknown. Chronic ketamine users (mostly ketamine abusers) may have structural and functional brain changes with associated memory problems. We are uncertain if this will occur at the frequency and duration proposed in this study.
- Bladder irritation and liver problems have been related to the repeated use of ketamine. We are uncertain if this will occur at the frequency and duration proposed in this study.
- The study treatment may also involve other risks, which are currently unforeseeable.
- If you become pregnant, the study treatment might involve risks to the embryo or fetus, which are currently unforeseeable.

### Clonidine Risks:

If you experience clinically significant elevated blood pressure (greater than 180 mmHg systolic blood pressure or greater than 105 mmHg diastolic blood pressure, or greater than 30 mmHg in systolic or diastolic blood pressure above baseline values), you will be treated with a blood pressure medication called clonidine. Clonidine will be given by mouth. Most common clonidine side effects include dry mouth (40 percent), drowsiness (33 percent), dizziness (16 percent), constipation (10 percent), sedation (10 percent), slow heart rate (4%), and low blood pressure. Syncope (or passing out) is a rare but possible side effect of clonidine.

### Ondansetron Risks:

If you experience clinically significant nausea which is causing discomfort and/or vomiting, you will be treated with an antiemetic medication called ondansetron. The most common side effects of ondansetron include constipation (10 percent) and headache.





Changing What's Possible


Version Date: 2/28/2023

## Alprazolam Risks:

If you experience clinically significant anxiety which is causing psychiatric distress or discomfort such as tense muscles, hyperventilation, or trembling, you will be treated with an anxiolytic medication called alprazolam. The most common side effects of alprazolam include drowsiness, decreased alertness, confusion, ataxia, memory impairment, and hypotension.

<u>Interviews and Surveys:</u> The questions that will be asked may be sensitive in nature and may make you feel uncomfortable. You may be asked personal questions that you find distressing. You may refuse to answer any question(s) that you do not wish to answer.

<u>Electrocardiogram (ECG)</u>: The ECG procedure may cause some mild discomfort during the placement and removal of the leads to and from the skin. You may also experience some local irritation, redness, or burning in the areas where the leads are attached.

## Risk of Loss of Confidentiality

There is a risk of a loss of confidentiality of your personal information as a result of participation in this study. Some answers you give during the research visits (like whether you use illegal drugs) may put you at risk if other people find out. To keep what you say private, your study records will use a code number instead of your name. We will protect your records to the extent allowed by law by keeping all your materials in locked file cabinets only accessible by research staff and all computer files will be secure password-protected files only accessed by research staff. Your research records are kept separate from your other medical records. Only research staff will have access to your private information.

# <u>Limits of Confidentiality</u>:

Suspected or known abuse or neglect of a child, disabled or elder abuse, or threatened violence to self or others may be reported to appropriate authorities.

<u>Unknown Risks:</u> The experimental treatments may have unknown side effects. The researchers will let you know if they learn anything during the course of the study that might make you change your mind about participating in the study.

### E. MEDICAL RECORDS AND/OR CERTIFICATE OF CONFIDENTIALITY

Information about your study participation will not be in your medical record. This means that neither your research participation nor any of your research results will be included in any MUSC medical record. This means that your research participation, saliva and pregnancy testing, and responses to questionnaires will not be included in your MUSC medical record.

## F. BENEFITS

If you receive ketamine, and it is more successful in treating your conditions compared to other standard treatments for smoking cessation, you may benefit from participating in the study. However, given the





Changing What's Possible


Version Date: 2/28/2023

investigational nature of this study, benefit cannot be guaranteed or promised. Information gained from this study may help other investigators have a better understanding of the treatment of tobacco use disorder.

### G. COSTS

There will be no cost to you because of participation in this study. If you choose to receive text message study reminders, normal data and usage rates will apply.

### H. PAYMENT TO PARTICIPANTS

Initial evaluation, three weekly medication sessions, and 2 follow up visits will not result in compensation other than reimbursement for time and local travel expenses. Reimbursement will be a flat rate of \$100 to cover compensation for time and travel for each in-person clinic visit. Payment for local travel expenses will be made using a prepaid debit card, called a ClinCard. It works like a bank debit card and you may use the card to purchase goods or services everywhere Debit MasterCard is accepted. You will be given a ClinCard at the beginning of the study. Each time you receive payment for participation in this study, the money will be added to the card, as outlined in the payment schedule above. Details of the debit card system are explained on an additional sheet. Payments that you receive from MUSC for participating in a research study are considered taxable income per IRS regulations. Payment types may include, but are not limited to: checks, cash, gift certificates/cards, personal property, and other items of value. If the total amount of payment you receive from MUSC reaches or exceeds \$600.00 in a calendar year, you will be issued a Form 1099.

#### I. ALTERNATIVES

If you choose not to participate in this study, you could receive other treatments for your condition. The standard therapies for tobacco use disorder include both medications (such as varenicline, bupropion, and nicotine replacement therapy) and counseling-based treatments (including group sessions such as individual or group counseling sessions).

# Withdrawal from the Study

Your participation in this study is voluntary. You may refuse to take part in or stop taking part in this study at any time. You should talk with the investigator in charge of this study. if you decide to do this. Your decision not to take part in the study will not affect your current or future medical care or any benefits to which you are entitled. The investigators and/or the sponsor may stop your participation in this study at any time if they decide it is in your best interest. They may also do this if you do not follow the investigator's instructions, or if the study is stopped by the study sponsor, the institutional review board (IRB), or by a regulatory agency (such as the FDA). If your participation is ended for medical reasons, you will be referred to a doctor or other health professional for care. You will be responsible for the cost of these services.




Version Date: 2/28/2023

#### J. DATA SHARING

Information about you (including your identifiable private information and/or any identifiable biospecimens) may have all of your identifiers removed and used for future research studies or distributed to other researchers for future research without additional informed consent from you or your legally authorized representative.

## **K. DISCLOSURE OF RESULTS**

Study data will not be shared with participants to maintain confidentiality.

# L. <u>AUTHORIZATION TO USE AND DISCLOSE (RELEASE) MEDICAL INFORMATION</u>

As part of this research study, your study doctor and his/her research team will keep records of your participation in this study.

The health information MUSC may use or disclose (release) for this research study includes information in your medical record, results of physical exams, medical history, lab tests or certain health information indicating or relating to your condition.

Your study doctor and his/her research team will use and disclose (release) your health information to conduct this study. The health information listed above may be used by and/or disclosed (released) to the following, as applicable:

- The sponsor of the study including its agents such as data repositories or contract research organizations monitoring the study;
- Other institutions and investigators participating in the study;
- Data Safety Monitoring Boards;
- Accrediting agencies;
- Clinical staff not involved in the study whom may become involved if it is relevant;
- Parents of minor children if less than 16 years old. Parents of children 16 years old or older require authorization from the child; or
- Health insurer or payer in order to secure payment for covered treatment;
- Federal and state agencies and MUSC committees having authority over the study such as:
  - The Institutional Review Board (IRB) overseeing this study; Committees with quality improvement responsibilities; Office of Human Research Protections; Food and Drug Administration; National Institutes of Health or Other governmental offices, such as a public health agency or as required by law.

Those persons who receive your health information may not be required by Federal privacy laws (such as the Privacy Rule) to protect it and may share your information with others without your permission, if permitted by laws governing them. You do not have to sign this consent form. If you choose not to sign, it will not affect your treatment, payment or enrollment in any health plan or affect






Version Date: 2/28/2023

your eligibility for benefits. However, you will not be allowed to be a participant in this research study.

You will be given a copy of this consent form. Your authorization will expire at the conclusion of this study or, if you are participating in a study designed for the development of a drug or device, your authorization will remain in effect until the drug or device is approved by the FDA or until the company's application to study the drug/device is withdrawn. You have the right to withdraw your agreement at any time. You can do this by giving written notice to your study doctor. If you withdraw your agreement, you will not be allowed to continue participation in this research study. However, the information that has already been collected will still be used and released as described above. You have the right to review your health information that is created during your participation in this study. After the study is completed, you may request this information.

Your health information will be used or disclosed when required by law. Your health information may be shared with a public health authority that is authorized by law to collect or receive such information for the purpose of preventing or controlling disease, injury or disability and for conducting public health surveillance, investigations or interventions. No publication or public presentation about the research study will reveal your identity without another signed authorization from you.

If you have questions or concerns about this Authorization or your privacy rights, please contact MUSC's Privacy Officer at (843) 792-8740.

Regulations require that you be given a copy of the MUSC Notice of Privacy Practices (NPP) describing the practices of MUSC regarding your health information. One can be found at the end of this form.

## M. SIGNIFICANT NEW FINDINGS

If there are significant new findings during the course of the study, you will be notified.

## N. STUDENT PARTICIPATION

Your participation or discontinuance will not constitute an element of your academic performance, nor will it be a part of your academic record at this Institution.

### O. EMPLOYEE PARTICIPATION

Your participation or discontinuance will not constitute an element of your job performance or evaluation, nor will it be a part of your personnel record at this Institution.

### P. CLINICAL TRIALS.GOV




Version Date: 2/28/2023

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Q. COLLECTION OF SPECIMENS

Saliva specimens will be collected in this study. All participants will provide a saliva sample during the screening phase and at each subsequent visit. Urine samples will be collected from individuals of childbearing potential to be checked for pregnancy at the baseline visit and every medication visit. Results of saliva and urine testing (pregnancy) will not be made a part of your medical record. These specimens will be used solely as part of this research study and will not be shared with other investigators or used for commercial profit. All specimens will be appropriately discarded with out identifying markers.

## **R. FUTURE CONTACT**

| The researcher in charge of this study might like to contact you in the future about other research opportunities. Please initial by your choice below: |
|---|
| Yes, I agree to be contacted |
| No, I do not agree to be contacted |
| You have the option of receiving appointment reminders and link to study surveys through tex messages for virtual follow-up visits. Should you elect to receive text messages, normal cellular data usage and rates will apply. Please initial by your choice below for paper consents, or scroll down to the bottom of the screen and select your choice electronically: |
| Yes, I agree to be contacted via text message |
| No, I do not agree to be contacted via text message |

Results of this research will be used for the purposes described in this study. This information may be published, but you will not be identified. Information that is obtained concerning this research that can be identified with you will remain confidential to the extent possible within State and Federal law. The sponsor and the Food and Drug Administration (FDA) will receive copies of the research records. The investigators associated with this study, employees of the sponsor, the FDA, and the MUSC Institutional Review Board for Human Research will have access to identifying information. All records in South Carolina are subject to subpoena by a court of law.

In the event of a study related injury, you should immediately go to the emergency room of the Medical University Hospital, or in case of an emergency go to the nearest hospital, and tell the physician on call that you are in a research study. They will call your study doctor who will make arrangements for your treatment. If the study sponsor does not pay for your treatment, the Medical University Hospital and the




Version Date: 2/28/2023

physicians who render treatment to you will bill your insurance company. If your insurance company denies coverage or insurance is not available, you will be responsible for payment for all services rendered to you.

Your participation in this study is voluntary. You may refuse to take part in or stop taking part in this study at any time. You should call the investigator in charge of this study if you decide to do this. The data collected on you to this point remains part of the study database and may not be removed. Your decision not to take part in the study will not affect your current or future medical care or any benefits to which you are entitled.

The investigators and/or the sponsor may stop your participation in this study at any time if they decide it is in your best interest. They may also do this if you do not follow the investigator's instructions.

## **Volunteers Statement**

I have been given a chance to ask questions about this research study. These questions have been answered to my satisfaction. If I have any more questions about my participation in this study or study related injury, I may contact the investigator in charge of the study (Dr. Emily Amador) at (843) 608-1216 or via e-mail at amador@musc.edu. I may contact the Medical University of SC Patient and Family Care Liaison (843) 792-5555 concerning medical treatment.

If I have any questions, problems, or concerns, desire further information or wish to offer input, I may contact the Medical University of SC Institutional Review Board for Human Research IRB Manager or the Office of Research Integrity Director at (843) 792-4148. This includes any questions about my rights as a research subject in this study.

I agree to participate in this study. I have been given a copy of this form for my own records. Please sign below for paper consents or scroll to the bottom of the screen to provide an electronic signature.

| Signature of Participant | Date |
|---------------------------------------|------|
| Printed Name of Participant | Date |
| Signature of Person Obtaining Consent | Date |

